CLINICAL TRIAL: NCT03311152
Title: Diagnostic Accuracy of the Circulating Cell-free DNA-based Epigenetic Biomarker MSEPT9 for Hepatocellular Carcinoma Detection Among Cirrhotic Patients: the SEPT9-CROSS Study
Brief Title: Circulating Cell-free DNA-based Epigenetic Biomarker MSEPT9 for Hepatocellular Carcinoma Detection in Cirrhosis
Acronym: SEPT9-CROSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Groupement Interrégional de Recherche Clinique et d'Innovation (Other); Epigenomics, Inc (Industry); New Day Diagnostics (Network)
Responsible Party: Principal Investigator, OUSSALAH Abderrahim, MD, PhD, OUSSALAH Abderrahim, MD, PhD, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2017-A01885-48
Record Dates: First submitted 2017-10-05; First posted 2017-10-17 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis
Keywords: Hepatocellular carcinoma; Cirrhosis; Circulating epigenetic biomarker; Plasma biomarker; SEPT9; Septin9; DNA methylation biomarker; Circulating DNA methylation biomarker; Alpha-fetoprotein
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Intervention Model Description: Cross-sectional
Who Masked: Participant, Care Provider, Investigator
Masking Description: The index test (mSEPT9) will be reported at the final step of the research, at time of data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCC-free cirrhotic patients (Controls) (Experimental): Cirrhotic patients enrolled in an HCC screening program by abdominal ultrasound and AFP every six months and followed at the Department of Hepatology of the University Hospital of Nancy. Each patient included will undergo a diagnostic test called "Epi proColon 2.0 CE" from Epigenomics, Inc (Berlin, Germany) also known as Plasma mSEPT9 test.
  Interventions: Diagnostic Test: "Epi proColon 2.0 CE" test from Epigenomics, Inc (Berlin, Germany)
- HCC-positive cirrhotic patients (Cases) (Experimental): Cirrhotic patients followed at the Department of Hepatology of the University Hospital of Nancy who presents an HCC according to the AASLD guidelines. Each patient included will undergo a diagnostic test called "Epi proColon 2.0 CE" from Epigenomics, Inc (Berlin, Germany) also known as Plasma mSEPT9 test.
  Interventions: Diagnostic Test: "Epi proColon 2.0 CE" test from Epigenomics, Inc (Berlin, Germany)

INTERVENTIONS:
Diagnostic Test: "Epi proColon 2.0 CE" test from Epigenomics, Inc (Berlin, Germany) — The mSEPT9 assay consists of DNA extraction from plasma, bisulfite conversion of DNA, purification of bis-DNA, and real-time PCR.
  Other Names: Plasma mSEPT9 test

SUMMARY:
Prospective evaluation of the circulating cell-free DNA-based epigenetic biomarker (mSEPT9) through a cross-sectional biomarker phase II design. The aim of the SEPT9-CROSS study is to assess the diagnostic accuracy of the plasma mSEPT9 biomarker in a large-scale study of 639 cirrhotic patients recruited in the participating centers.

DETAILED DESCRIPTION:
Epigenetic alterations are a common hallmark of human cancer. Single epigenetic markers are starting to be incorporated into clinical practice; however, the translational use of these biomarkers has not been validated at the 'omics' level. This is strikingly the case in hepatocellular carcinoma (HCC) which represent the most common primary malignant tumor of the liver. Alpha-fetoprotein (AFP) has been widely used as a diagnostic marker of HCC; however, according to international guidelines (AASLD, EASL), AFP is unsufﬁciently sensitive or unsufﬁciently speciﬁc for use in a screening assay. Aberrantly methylated DNA sequences frequently occur in tumors and are detected in the circulation of cancer patients by polymerase chain reaction (PCR). SEPT9 is a significant epi-driver gene in liver carcinogenesis. The SEPT9 gene is a key regulator of cell division and tumor suppressor whose hypermethylation is associated with carcinogenesis. SEPT9 is involved in the onset of rat hepatocarcinogenesis and SEPT9-promoter hypermethylation was reported in HCC in man. SEPT9 expression is turned on in cells throughout the body and absent or diminished by aberrant promoter methylation in several types of cancer. Through an initial proof-of-concept pilot study from France and an independent replication study from Germany, we showed that the circulating cell-free DNA methylation-based epigenetic biomarker mSEPT9 is a promising plasma biomarker for diagnosing HCC in cirrhotic patients. The aim of the SEPT9-CROSS study is to confirm the diagnostic accuracy of the biomarker in a large-scale study of 630 cirrhotic patients recruited in the participating centers.

ELIGIBILITY:
INCLUSION CRITERIA

* Patient aged 18 and over.
* Patient with a diagnosis of cirrhosis (alcohol, HBV, HBC, NASH, hemochromatosis, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis) with or without hepatocellular carcinoma (for each arm).
* Affiliation to the French Social Security System (Health Insurance)

NON-INCLUSION CRITERIA FOR CASES :

* Malignant liver tumor other than HCC: cholangiocarcinoma, hepatic metastasis of a carcinoma (e.g., colorectal adenocarcinoma);
* History of HCC treated by surgical resection, focal destruction [radiofrequency, stereotactic radiotherapy (CYBERKNIFE®)], arterial chemoembolization, or radioembolization within the last five years.

NON-INCLUSION CRITERIA FOR CASES AND CONTROLS:

* Legal protection measures;
* Pregnant woman;
* Hemodialysis, ongoing (possibility of interference with the test);
* Presence of associated cancer (e.g., colorectal adenocarcinoma, urothelial carcinoma, breast carcinoma, etc.) since less than five years;
* Presence of a hematological malignancy (no time limit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Presence of hepatocellular carcinoma. | The diagnosis of HCC will be based on overall patient's evaluation including clinical, biological and imaging workup which will be carried out during the consultation and/or the three months preceding or following the inclusion consultation.
  The diagnosis of hepatocellular carcinoma will be based on the guidelines of the American Association for the Study of Liver Diseases (AASLD) (Hepatology. 2011;53:1020-2). The adjudicating physicians will be blinded to patient results associated with the mSEPT9 test.

SECONDARY OUTCOMES:
Presence of early hepatocellular carcinoma. Early hepatocellular carcinoma will be defined as a tumor smaller than 30 mm according to Kudo M (Liver Cancer. 2013;2:69-72). | The diagnosis will be based on an overall patient's evaluation including clinical, biological and imaging workup which will be carried out during the consultation and/or the three months preceding or following the inclusion consultation.
  The diagnosis of hepatocellular carcinoma will be based on the guidelines of the American Association for the Study of Liver Diseases (AASLD) (Hepatology. 2011;53:1020-2). The adjudicating physicians will be blinded to patient results associated with the mSEPT9 test.

CONTACTS AND LOCATIONS:
Overall Officials: Abderrahim OUSSALAH, MD, PhD, Principal Investigator — University Hospital of Nancy, INSERM UMR_S 1256, Faculty of Medicine of Nancy, University of Lorraine
Locations (1):
- University Hospital of Nancy (CHRU de Nancy), Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
Final report, publication in a peer review journal. Main data and supplemental data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Final report after data completion.
Access Criteria: After the publication of study results.